CLINICAL TRIAL: NCT04024787
Title: Neural Responses and Connectivity During Rest, Memory Encoding and Emotional Stimulation in Chronic Insomnia, and Their Relationships With Insomnia Treatment: a Wait-list Controlled Randomized Trial of Cognitive-behavioural Therapy for Insomnia
Brief Title: Impact of Insomnia Treatment on Brain Responses During Resting-state and Cognitive Tasks
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Concordia University, Montreal (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Thanh Dang-Vu, Principal Investigator, Associate Professor, Concordia University, Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 30011416
Record Dates: First submitted 2019-07-12; First posted 2019-07-18 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Chronic Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial. Participants with chronic insomnia are randomized to either immediate cognitive-behavioural therapy or a 3-month wait-list period using a 1:1 allocation ratio. Randomization is conducted with block sizes of 4 participants. Randomization results are contained in sealed opaque envelopes that are opened in the presence of the participants after the completion of the pre-treatment assessment. A second assessment will be conducted after the treatment or waiting period. A follow-up assessment is conducted 12 months after the completion of the post-treatment assessment. A group of good sleepers, matched on age and gender with the insomniacs, will also be recruited and assessed at baseline only to provide a normative reference group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate intervention (Experimental)
  Interventions: Behavioral: Cognitive-Behavioural therapy for insomnia (CBT-I)
- Waitlist (No Intervention)

INTERVENTIONS:
Behavioral: Cognitive-Behavioural therapy for insomnia (CBT-I) — Participants with chronic primary insomnia are randomized into 2 groups with a 1:1 allocation ratio, after the completion of the pre-treatment assessment. Post-treatment and post-waitlist assessment occur after the 3-month treatment or waiting period.
  One group will receive the intervention immediately after the pre-treatment assessment and the other group will receive the intervention after a waiting period of 3 months. The intervention consists of manualized cognitive-behavioural therapy for insomnia. This treatment includes psychoeducation about sleep and circadian rhythms, stimulus control, sleep restriction, relaxation, and cognitive therapy. The therapy is administered individually. Participants meet for 8 sessions of 50 minutes spread over 12 weeks.
  Arms: Immediate intervention

SUMMARY:
Individuals with chronic insomnia have persistent difficulty falling and staying asleep, as well as complaints of altered daytime functioning that may be associated with cognitive impairments. The neural processes underlying these daytime complaints may involve abnormal activation of brain regions and neural networks involved in working memory, memory encoding and emotions. The goal of this study is to assess whether a psychological treatment for insomnia will reverse these abnormalities in brain responses to cognitive tasks and at rest. A secondary objective of the study is to characterize impairments in attentional processing and assess if the impairments can be reversed by the psychological treatment. We hypothesized that the psychological treatment for insomnia will lead to a normalization of the brain responses to working memory, declarative memory encoding, insomnia-related stimuli, and the functional connectivity within the default-mode and limbic networks.

DETAILED DESCRIPTION:
Study hypothesis

Brain responses associated with working memory task and declarative memory encoding will be decreased in chronic insomnia compared to good sleepers and, among individuals with chronic insomnia, cognitive-behavioral therapy for insomnia will lead to larger recovery in these brain responses, compared to a 3-month wait period.

Brain responses to emotional stimulation, especially to insomnia-related stimuli, will be increased in chronic insomnia compared to good sleepers, and, among individuals with chronic insomnia, cognitive-behavioral therapy for insomnia will lead to larger reduction in these brain responses, compared to a 3-month wait period.

Connectivity in the default-mode and limbic networks during resting-state will be increased in chronic insomnia compared to good sleepers, and, among individuals with chronic insomnia, cognitive-behavioral therapy for insomnia will lead to larger reduction in this connectivity, compared to a 3-month wait period.

ELIGIBILITY:
Inclusion Criteria:

80 participants with chronic primary insomnia (40 per group) 40 good sleepers

Exclusion Criteria:

1. Older than 65 y.o. or younger than 25 y.o.
2. Contraindication to the MRI scanning
3. Current neurological disorder
4. Past history of brain lesion
5. Major surgery (i.e., requiring general anesthesia) in the past 3 months
6. Untreated thyroid disorder
7. Chronic pain syndrome self-reported as interfering with sleep
8. Recent and severe infection in the past 3 months
9. Active cancer, or remitted cancer with cancer treatment within the last 2 years
10. Stroke
11. Myocardial infarct
12. Arterial bypass or angioplasty
13. Pacemaker
14. Heart failure causing limitation of ordinary physical activity
15. Renal insufficiency
16. Sleep apnea with an apnea-hypopnea index > 5/h
17. Restless legs syndrome with symptoms 3 days or more per week
18. Periodic limb movements during sleep with index > 15/h
19. REM-sleep behavior disorder
20. Narcolepsy and other central disorders of hypersomnolence
21. Sleepwalking more than once/month
22. Having worked on night shifts or rotating shifts for more than 2 weeks in the last 3 months or expecting to do so during the study period
23. Severe mental disorders: bipolar disorder (Type I), schizophrenia, anxiety disorders, major depressive disorder, current substance use disorder, current post-traumatic stress disorder
24. Current suicidality
25. Frequent alcohol consumption (>10 glasses/week) or use of cannabis (more than once a week) or illicit drugs (more than once a month)
26. Smoking cigarettes more than 10 cigarettes/day
27. Pregnant or breastfeeding women
28. Current psychotherapy or past cognitive-behavioural therapy for insomnia
29. Current use of medication for depression or anxiety
30. Unable to stop hypnosedative medications for at least 2 weeks prior to the first assessment
31. For good sleepers: insomnia symptoms more than 3 times/ week.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-07-30 (Actual); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Functional magnetic resonance imaging (fMRI) to examine brain responses to working memory with increasing task difficulty | 3 months
  Functional magnetic resonance imaging (fMRI) will be used to look at changes in brain activations to working memory in individuals with chronic insomnia compared to good sleepers, as well as the modifications in these brain activations after cognitive-behavioral therapy for insomnia.
Functional magnetic resonance imaging (fMRI) to examine brain responses to declarative memory encoding | 3 months
  Functional magnetic resonance imaging (fMRI) will be used to look at changes in brain activations to declarative memory encoding in individuals with chronic insomnia compared to good sleepers, as well as the modifications in these brain activations after cognitive-behavioral therapy for insomnia.
Functional magnetic resonance imaging (fMRI) to examine brain responses to insomnia-related stimuli | 3 months
  Functional magnetic resonance imaging (fMRI) will be used to look at changes in brain activations to insomnia-related pictures in individuals with chronic insomnia compared to good sleepers, as well as the modifications in these brain activations after cognitive-behavioral therapy for insomnia.
Functional magnetic resonance imaging (fMRI) to examine functional connectivity within the default-mode and limbic networks at rest | 3 months
  Functional magnetic resonance imaging (fMRI) will be used to look at changes in resting state functional connectivity in individuals with chronic insomnia compared to good sleepers, as well as the modifications in this functional connectivity after cognitive-behavioral therapy for insomnia, with a focus on the default-mode and limbic networks.

SECONDARY OUTCOMES:
Insomnia Severity Index (ISI) | 3 months and 1 year
  Self-reported insomnia severity
Pittsburgh Sleep Quality Index (PSQI) | 3 months and 1 year
  Self-reported sleep quality
Total sleep time | 3 months and 1 year
  Self-reported total sleep time from 14-day sleep diary
Total sleep time | 3 months
  Total sleep time from 14-day actigraphy
Sleep latency | 3 months and 1 year
  Self-reported sleep latency from 14-day sleep diary
Sleep latency | 3 months
  Sleep latency from 14-day actigraphy
Wake-after-sleep-onset (WASO) | 3 months and 1 year
  Self-reported duration of wake-after-sleep-onset from 14-day sleep diary
Wake-after-sleep-onset (WASO) | 3 months
  Duration of wake-after-sleep-onset from 14-day actigraphy
Sleep efficiency | 3 months and 1 year
  Self-reported sleep efficiency from 14-day sleep diary
Sleep efficiency | 3 months
  Sleep efficiency from 14-day actigraphy
Diagnosis of insomnia disorder | 3 months and 1 year
  A trained interviewer evaluates the presence of an insomnia disorder using the SCID-V
PSG total sleep time | 3 months
  Total sleep time from overnight polysomnography
PSG sleep latency | 3 months
  Sleep latency from overnight polysomnography
PSG wake-after-sleep-onset (WASO) | 3 months
  Duration of wake-after-sleep-onset from overnight polysomnography
PSG sleep efficiency | 3 months
  Sleep efficiency from overnight polysomnography
Sleep stage durations (N1, N2, N3, REM) | 3 months
  Durations of each sleep stage from overnight polysomnography
Arousal index | 3 months
  Number of EEG arousals per hour from overnight polysomnography
Spindle density | 3 months
  Number of sleep spindles per minute of stage N2-N3 sleep from overnight polysomnography
Dim light melatonin onset (DLMO) | 3 months
  Objective measure of central circadian timing (dim light melatonin onset; DLMO) will be obtained from hourly evening saliva samples
Cortisol | 3 months
  Cortisol will be assessed using salivary samples collected at bedtime, awakening and 45 minutes after awakening
Heart rate variability | 3 months
  Heart rate variability will be measured using the electrocardiogram leads during the overnight assessments
Blood pressure | 3 months
  Blood pressure is assessed using an oscillometer measurement of systolic and diastolic blood pressure in the morning following the overnight assessments
Circulating interleukin-6 | 3 months
  Markers will be quantified using blood sample during the overnight assessments
Circulating tumor necrosis factor-alpha | 3 months
  Markers will be quantified using blood sample during the overnight assessments
Circulating C-reactive protein | 3 months
  Markers will be quantified using blood sample during the overnight assessments
Circulating neurotrophic factor BDNF | 3 months
  Markers will be quantified using blood sample during the overnight assessments
Beck Depression Inventory (BDI) | 3 months and 1 year
State-Trait Inventory for Cognitive and Somatic Anxiety (STICSA) | 3 months and 1 year
Sahlgrenska Academy Self-reported Cognitive Impairment Questionnaire (SASCI-Q, adapted version) | 3 months and 1 year
  Questionnaire assessing self-reported (subjective) memory complaints. Total score ranges from 29 to 203 (higher score reflects more self-reported cognitive complaints).
Work and Social Adjustment Scale (WSAS) | 3 months and 1 year
  Self-reported measure assessing perceived functional impairment associated with insomnia. Total score ranges from 0 to 40 (lower score reflects less impairment).
The Implicit Positive and Negative Affect Test (IPANAT) | 3 months and 1 year
Beliefs and Attitudes about Sleep (DBAS) | 3 months and 1 year
Daytime Insomnia Symptom Response Scale (DISRS) | 3 months and 1 year
  Self-report measures assessing sleep-related rumination
Attention | 3 months
  Attention will be assessed using computerized divided attention and multitasking tasks assessed in the evening and morning of the overnight assessments
Gray matter volume (GMV) | 3 months
  Brain morphometric measure from MRI
Cortical thickness | 3 months
  Brain morphometric measure from MRI
White matter integrity (fractional anisotropy, mean diffusivity) | 3 months
  Brain measure from MRI
GABA | 3 months
  GABA concentration from Magnetic Resonance Spectroscopy (in the anterior cingulate cortex)
Trier Inventory for Chronic Stress - short form | 3 months and 1 year
Subjective happiness scale | 3 months and 1 year
  Self-reported measure of global subjective happiness. Total score ranges from 4 to 28 (higher score reflects greater happiness).
Temporal experience of pleasure scale (adapted version) | 3 months and 1 year
  Self-reported measure of anticipatory and consummatory facets of pleasure. Total score ranges from 18 to 52 (higher score reflects greater pleasure).
Fatigue symptom inventory | 3 months and 1 year
Positive and Negative Affect Schedule | 3 months and 1 year
Munich Chronotype Questionnaire (MCTQ) | 3 months and 1 year
  Questionnaire on self-reported sleep habits, assessing individual chronotype (e.g., early type, normal type late type).

CONTACTS AND LOCATIONS:
Overall Officials: Thanh Dang-Vu, MD PhD, Principal Investigator — Concordia University, Montreal
Locations (1):
- Perform Center, Concordia University, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No